CLINICAL TRIAL: NCT04370470
Title: Development of Assessments for Later Stage Huntington's Disease: UHDRS Structured Interview of Function and HD Clinical Status Questionnaire
Brief Title: Development of Assessments for Later Stage HD
Acronym: LSA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: C-000619
Record Dates: First submitted 2020-04-24; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-01

CONDITIONS: Huntington Disease
Keywords: CHDI; Huntington Disease; Huntington's Disease; Huntington's Disease Later Stage
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Later Stage HD Assessments (LSA) is an observational, multinational study aiming at developing two assessments that can be used to measure critical milestones and events during the later stages of Huntington's disease (HD). An important aspect of the evaluation will be to assess whether the assessments can be administered to a companion either in-person or remotely (i.e. by phone contact with the companion). Therefore, these assessments will be evaluated for their internal consistency, reliability and validity. Once established, these assessments may be incorporated into a large scale, global observational study of HD and/or other HD clinical studies as well as use them for planning clinical trials.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the internal consistency, reliability and validity of two assessments: (1) UHDRS Structured Interview of Function (SIF) that incorporates the UHDRS Total Functional Capacity, Functional Assessment Scale, and Independence Scale (UHDRS TFC, FAS and IS), and (2) the HD Clinical Status Questionnaire (HDCSQ). There will be two study parts: Part 1 will measure the performance of the UHDRS SIF assessment compared to the original UHDRS TFC, FAS and IS using a cross-over design by collecting data from the Manifest HD gene expansion carrier participants (Manifest HDGEC Participants) and their companions (Companion Participants) via an in-person baseline visit and a follow-up visit by phone. Part 2 will assess the UHDRS SIF and the HDCSQ using a cross-sectional design by collecting data from the Companion Participants via a follow-up visit by phone. Participants of Part 1 are eligible to participate in Part 2.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following inclusion criteria to participate in this study:

All Participants

1. Individual of either gender
2. Fluent in English
3. Must be willing and able to provide informed consent or have a legal representative willing and able to provide assent

Manifest HDGEC Participants

1. Must be an active participant in the Enroll-HD study. An active participant is defined as a participant who has successfully enrolled in the Enroll-HD study and completed the Enroll-HD study baseline visit.
2. Age≥20 years
3. CAG repeat length≥36
4. DCL=4
5. Inclusion score of 16 at the time of the participant's most recent Enroll-HD study visit (for inclusion score calculation, see Appendix A - Inclusion Score Calculation) Companion Participants

1. Age≥18 years 2. A person who, in his/her opinion, has sufficient interface and knowledge of the Manifest HDGEC Participant's capabilities and daily activities 3. Acceptable to the Manifest HDGEC Participant and the Site Investigator or the Site Investigator's designees

Exclusion Criteria:

People who meet the following criteria will be excluded from participating in this study:

1. Individuals with choreic movement disorders in the context of a laboratory verified non-expansion mutation for the Huntingtin gene
2. Manifest HDGEC Participants with Juvenile-onset HD (rater estimate of age of onset <20 years old)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Manifest HDGEC Participants: Manifest HDGEC Participants must be participants in the Enroll-HD study. Manifest HDGEC Participants will be recruited from English-speaking study sites participating in the Enroll-HD study.
  Companion Participants: Companions Participants will be identified for Manifest HDGEC Participants and asked to participate. A Companion Participant's participation for a Manifest HDGEC participant is mandatory.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The UHDRS SIF ratings | 3 weeks
  The equivalence of the original UHDRS function scales (TFC, FAS and IS) and the UHDRS SIF will be evaluated using a cross-over design study, with two baseline measurements and one follow up measurement. We will use ICC (Intraclass Correlation Coefficient) and Lin's correlation coefficient will be used to measure the agreement between raters across Participants.
Clinimetric properties of the UHDRS SIF | 3 weeks
  To assess the clinimetric properties of the UHDRS SIF we will use Classical Test Theory (CTT) and Item Response Theory (IRT)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (9):
  - The Board of Trustees of the University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Regents of the University of California, San Diego, La Jolla, California
  - Regents of the University of California, Los Angeles, Los Angeles, California
  - Rocky Mountain Movement Disorders Center, P.C, Englewood, Colorado
  - Rush Universiity Medical Center, Chicago, Illinois
  - Hereditary Neurological Disease Centre, Inc., Wichita, Kansas
  - Washington University, St Louis, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington
- United Kingdom (11):
  - The Chancellor, Masters and Scholars of the University of Cambridge, Cambridge, Cambridgeshire
  - Cardiff University, Wales, Cardiff
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Poole Hospital NHS, Poole, Dorset
  - Leicestershire Partnership NHS Trust, Leicester, Leicestershire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Leicester
  - Northumberland, Tyne &Wear NHS Foundation Trust of St. Nicholas Hospital, Newcastle upon Tyne, Tyne & Wear
  - Birmingham and Solihull Mental Health NHS Foundation, Birmingham, West Midlands
  - Leeds Teaching Hospitals NHS Trust, Leeds, Yorkshire
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Sheffield Children's NHS Foundation Trust, Sheffield